CLINICAL TRIAL: NCT04060420
Title: Yathu Yathu ("For us, by us"): A Cluster-randomized Trial of Comprehensive Community-based Peer-led Sexual and Reproductive Health Services for Adolescents and Young People Aged 15 to 24 in Lusaka, Zambia
Brief Title: Yathu Yathu: An Impact Evaluation of Community-based Peer-led Sexual and Reproductive Health Services
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Zambart (Other); Imperial College London (Other); Medical Research Council (funder; grant number: MR/R022216/1) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17104
Record Dates: First submitted 2019-08-12; First posted 2019-08-19 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases | interventions — Reproductive Health Services

STUDY DESIGN:
Intervention Model Description: This study is a cluster-randomised trial, with a total of 20 clusters across two communities (10 clusters per community). Within each community, these 10 clusters have been randomised to intervention or control arm using restricted randomisation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive sexual and reproductive health services (Experimental): In clusters randomised to the Yathu Yathu intervention, the comprehensive, community-based and peer-led intervention is being delivered. In addition to delivery of sexual and reproductive health services through community-based hubs, the intervention includes the Yathu Yathu prevention points cards, with which adolescents and young people can accrue points for accessing services at the Yathu Yathu hub and local health facility, and redeem rewards using these points.
  Interventions: Other: Comprehensive sexual and reproductive health services
- Standard of care (No Intervention): In the comparison arm, adolescents and young people will have access to sexual and reproductive health services at the local health facility. They will also have a Yathu Yathu prevention points card, with which they can accrue points for accessing sexual and reproductive health services at the local health facility and redeem rewards using these points.

INTERVENTIONS:
Other: Comprehensive sexual and reproductive health services — The intervention includes community-based and peer-led delivery of comprehensive sexual and reproductive health services and a Yathu Yathu prevention points card, which is a card that adolescents and young people can use to gain points for accessing services and use these points to redeem rewards.
  Arms: Comprehensive sexual and reproductive health services

SUMMARY:
This trial evaluates the impact of providing comprehensive, community-based and peer-led sexual and reproductive health services to adolescents and young people aged 15 to 24 on their knowledge of their HIV status. The trial includes 20 clusters in two communities, half the clusters receive the intervention. After 18-months of implementation, a cross-sectional survey will be conducted to evaluate the impact of the intervention on the primary outcome: knowledge of HIV status.

DETAILED DESCRIPTION:
Through a cluster-randomised trial, this study will address the research question: Do community-based peer-led interventions increase knowledge of HIV status and coverage of sexual and reproductive health services among adolescents and young people in Lusaka, Zambia, compared to current standard of care? To address this question, the study aims to build a rigorous evidence-base of the effectiveness of community-based, peer-led HIV services designed with and for adolescents and young people living in Lusaka, Zambia, and evidence of the process of delivering such an intervention to support replication and scale-up if the intervention is effective.

The intervention, called Yathu Yathu (For us, by us), was designed with adolescents and young people in a formative research study. The Yathu Yathu intervention includes: 1) delivery of comprehensive sexual and reproductive health services by peer support workers, lay counsellors and a nurse at community-based hubs, and 2) an innovative "prevention points card" system. The prevention points cards are intended to incentivise service use by allowing adolescents and young people to accrue points for accessing services and redeem rewards using these points. At the start of the intervention period, trained enumerators will systematically visit and enumerate all households in the 20 study clusters. For household members aged 15 to 24, the enumerators will offer the individual a prevention points card. A third component is mobile phone-based support groups. These groups will initially be set-up among HIV-positive pregnant women, as a means to offer psychosocial support, with expansion of this portion of the intervention to other groups planned.

To evaluate the impact of the Yathu Yathu intervention, a cross-sectional survey among a random sample of approximately 2000 adolescents and young people will be conducted 18-months after implementation of the intervention. An embedded mixed-method process evaluation will provide evidence of service acceptability, feasibility, and of adolescents and young people's experiences with services. An economic evaluation will provide evidence of the costs and cost-effectiveness of the intervention package. Through these methods, this study will provide a rigorous and comprehensive evidence-base of whether Yathu Yathu can increase adolescents and young people access to sexual and reproductive health services, thereby contributing to their health and well-being.

ELIGIBILITY:
Inclusion Criteria for the cross-sectional survey to be conducted 18 months after implementation of the Yathu Yathu intervention:

* 16 - 26 years of age at time of the survey (15 to 24 at the time of household enumeration and distribution of the Yathu Yathu prevention points card)
* Residing within the cluster during enumeration of the cluster
* Received a prevention points card at the time of household enumeration
* Able and willing to provide informed consent.

Exclusion Criteria:

* Anything that, in the opinion of the investigator, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge of HIV status | Outcome measured at single time point, but refers to previous 1 year period.
  Defined as self-reported HIV positive status or reporting an HIV-test within the previous 1 year period.

SECONDARY OUTCOMES:
Coverage of sexual and reproductive health services | Outcome measured at single time point, but refers to the previous 1 year period.
  The average number of services accessed at least once the previous 1 year period.
Uptake of medical male circumcision services | Outcome measured at single time point, but refers to the previous 1 year period.
  Proportion of adolescent boys and young men accessing voluntary medical male circumcision services
Met need for family planning | Outcome measured at single time point, but refers to the previous 1 year period.
  Proportion of young women with met needs for family planning services
PrEP uptake and adherence | Outcome measured at single time point, but refers to the previous 1 year period.
  Self-reported uptake of and adherence to PrEP among individuals who are HIV negative
ART use | Outcome measured at single time point, but refers to the previous 1 year period.
  Self-reported current use of and retention on ART among individuals who are HIV positive
Pregnancies among young women | Outcome measured at single time point, but refers to the previous 1 year period.
  Proportion of young women reporting pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Helen Ayles, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Zambart, Lusaka, Zambia

REFERENCES:
- [Derived] Rotsaert A, Phiri M, Sigande L, Schaap A, Zulu-Phiri R, Simuyaba M, Mwape L, Floyd S, Fidler S, Hayes R, Simwinga M, Ayles H, Hensen B. Unmet need for contraceptives and unintended pregnancies among adolescent girls and young women aged 15 to 24 in Zambia: insights from the Yathu Yathu trial. Reprod Health. 2025 Nov 12;22(1):229. doi: 10.1186/s12978-025-02202-y. PMID 41225474
- [Derived] Phiri MM, Schaap A, Hensen B, Sigande L, Simuyaba M, Mwenge L, Zulu-Phiri R, Mwape L, Floyd S, Fidler S, Hayes R, Simwinga M, Ayles H. The impact of an innovative community-based peer-led intervention on uptake and coverage of sexual and reproductive health services among adolescents and young people 15-24 years old: results from the Yathu Yathu cluster randomised trial. BMC Public Health. 2024 May 28;24(1):1424. doi: 10.1186/s12889-024-18894-z. PMID 38807091
- [Derived] Hensen B, Phiri MM, Sigande L, Schaap A, Simuyaba M, Zulu-Phiri R, Mwape L, Floyd S, Fidler S, Hayes R, Simwinga M, Ayles H. Self-reported uptake of STI testing services among adolescents and young people aged 15-24 years: Findings from the Yathu Yathu cluster randomized trial in Lusaka, Zambia. PLOS Glob Public Health. 2024 Mar 4;4(3):e0002491. doi: 10.1371/journal.pgph.0002491. eCollection 2024. PMID 38437238
- [Derived] Hensen B, Floyd S, Phiri MM, Schaap A, Sigande L, Simuyaba M, Mwenge L, Zulu-Phiri R, Mwape L, Fidler S, Hayes R, Simwinga M, Ayles H. The impact of community-based, peer-led sexual and reproductive health services on knowledge of HIV status among adolescents and young people aged 15 to 24 in Lusaka, Zambia: The Yathu Yathu cluster-randomised trial. PLoS Med. 2023 Apr 21;20(4):e1004203. doi: 10.1371/journal.pmed.1004203. eCollection 2023 Apr. PMID 37083700
- [Derived] Phiri MM, Hensen B, Schaap A, Sigande L, Simuyaba M, Simwinga M, Floyd S, Fidler S, Hayes R, Ayles H. Adapting community-based sexual and reproductive health services for adolescents and young people aged 15-24 years in response to COVID-19 in Lusaka, Zambia: the implications on the uptake of HIV testing services. BMC Health Serv Res. 2022 Apr 14;22(1):503. doi: 10.1186/s12913-022-07878-7. PMID 35421966
- [Derived] Simuyaba M, Hensen B, Phiri M, Mwansa C, Mwenge L, Kabumbu M, Belemu S, Shanaube K, Schaap A, Floyd S, Fidler S, Hayes R, Ayles H, Simwinga M. Engaging young people in the design of a sexual reproductive health intervention: Lessons learnt from the Yathu Yathu ("For us, by us") formative study in Zambia. BMC Health Serv Res. 2021 Jul 29;21(1):753. doi: 10.1186/s12913-021-06696-7. PMID 34325696